CLINICAL TRIAL: NCT02108431
Title: Superior Postoperative Patient Comfort in Suprapubic Drainage Versus Transurethral Catheterization Following Robot-assisted Radical Prostatectomy: A Prospective Randomized Clinical Trial
Brief Title: Prospective Randomized Trial Comparing Urinary Diversion After Robot-assisted Radical Prostatectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Antonius Hospital Gronau (Other)
Responsible Party: Principal Investigator, J.H. Witt, MD., St. Antonius Hospital Gronau
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: U1111-1155-1458
Record Dates: First submitted 2014-03-31; First posted 2014-04-09 (Estimated); Last update posted 2014-04-09 (Estimated); Status verified 2014-04

CONDITIONS: Prostate Cancer
Keywords: urinary diversion; urethral catheter; suprapubic tube; radical prostatectomy; robotic surgery; discomfort; pain
MeSH Terms: conditions — Prostatic Neoplasms; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- balloon catheter for transurethral bladder-drainage (Experimental): intraoperatively placement of transurethral catheter after robot-assisted radical prostatectomy
  Interventions: Device: balloon catheter for transurethral bladder-drainage
- balloon catheter for suprapubic bladder-drainage (Active Comparator): intraoperatively placement of suprapubic catheter after robot-assisted radical prostatectomy
  Interventions: Device: balloon catheter for suprapubic bladder-drainage

INTERVENTIONS:
Device: balloon catheter for suprapubic bladder-drainage — suprapubic tube removal was allowed when the anastomosis was watertight, Day 5
  Other Names: UROMED; suprapubic tube; suprapubic device
  Arms: balloon catheter for suprapubic bladder-drainage
Device: balloon catheter for transurethral bladder-drainage — transurethral catheter withdrawal was allowed when the anastomosis was watertight, Day 5
  Other Names: UROMED
  Arms: balloon catheter for transurethral bladder-drainage

SUMMARY:
The purpose of the study is to determine, whether the urinary diversion via suprapubic cystostomy compared to transurethral catheterization after robot-assisted radical prostatectomy superior the postoperative patient comfort and reduce the postoperative bacteriuria.

ELIGIBILITY:
Inclusion Criteria:

1. Minimum age of 18 Years
2. Voluntarily agreement to participate in this study
3. Written informed-consent
4. Release of medical records for regulatory or research purposes
5. Clinically organ-confined prostate cancer

Exclusion Criteria:

1. BMI >40
2. History of catheterization
3. History of radiation
4. History of chemotherapy
5. Person's participating in any other research
6. Unable to provide informed consent

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2013-02; Primary Completion 2013-10 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Change of postoperative pain related to urinary drainage objectified by numeric rating scale (NRS) questionnaire within 5 days | postoperatively on day 1, 2, 3, 4 and 5 in the morning, at noon and in the evening
  To analyse the development of the postoperative pain related to urinary drainage patients completed NRS questionnaire three times a day: in the morning, at noon and in the evening until discharge of the catheter (regular 5 days after the surgery)

SECONDARY OUTCOMES:
Number of patients with bacteriuria | 5th day after the surgery
  Second void urine sample after catheter removal

CONTACTS AND LOCATIONS:
Overall Officials: Jawid Habibzada, MD., Study Chair — St. Antonius Hospital Gronau; Michael Godes, MD., Study Chair — St. Antonius Hospital Gronau
Locations (1):
- Department of Urology, Pediatric Urology and Urologic Oncology; St. Antonius-Hospital Gronau GmbH, Gronau, Germany